CLINICAL TRIAL: NCT01532076
Title: Effectiveness of Adipose Tissue Derived Mesenchymal Stem Cells as Osteogenic Component in Composite Grafts Versus Acellular Bone Graft Substitutes for Augmentation in the Treatment of Proximal Humeral Fractures as Model for Fractures of Osteoporotic Bone - a Prospective Randomized First in Men Proof of Principle Trial
Brief Title: Effectiveness of Adipose Tissue Derived Mesenchymal Stem Cells as Osteogenic Component in Composite Grafts
Acronym: ROBUST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 348/10
Record Dates: First submitted 2012-01-05; First posted 2012-02-13 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Osteoporotic Fractures
Keywords: osteoporosis; prox. humeral fracture; geriatric trauma; mesenchymal stem cells
MeSH Terms: conditions — Osteoporotic Fractures; Osteoporosis | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cellularized composite graft augmentation (Experimental): lipoaspiration by experienced plastic surgeon, isolation of SVF cells using a Cellution/CR800® cell isolation device and single use kits (Cytori Therapeutics Inc., San Diego) during open reduction and internal fixation, augmentation of bone with cell-seeded bone graft substitute;
  Interventions: Procedure: Cellularized composite graft augmentation
- Control acellular composite graft augmentation (Active Comparator): open reduction internal fixation (ORIF) of the fracture, augmentation with acellular bone graft substitute.
  Interventions: Procedure: Acellular composite graft augmentation

INTERVENTIONS:
Procedure: Cellularized composite graft augmentation — liposuction, cell isolation, embedding of SVF cells in fibrin gel, wrapping around hydroxyapatite granules
  Other Names: Cellution/CR800, Cytori, US; Tisseel, Baxter, Germany; Actifuse Microgranules, Apatech, Germany
  Arms: cellularized composite graft augmentation
Procedure: Acellular composite graft augmentation — Open reduction and internal fixation using acellular augmentation with fibrin embedded granulated hydroxyapatite
  Other Names: Tisseel, Baxter, Germany; Actifuse Microgranules, Apatech, Germany
  Arms: Control acellular composite graft augmentation

SUMMARY:
Failure rates of up to 30% are reported after proximal humeral fractures despite angular-stable devices. This may devastate not only the functional outcome but also the independence of elderly patients.

To increase bone mineral density and thereby holding-strength augmentation is an option. Autologous bone-graft, as current gold-standard, though is questionable in osteoporosis since osteoprogenitors are dysfunctional and the harvesting-morbidity considerable. Adipose tissue seems an alternative cell-source even in presence of osteoporosis.

Stromal vascular fraction (SVF) cells isolated from lipoaspirates display osteogenic and vasculogenic potential and can be harvested in high numbers. Expansion associated with costly good-manufacturers-practice facilities is avoidable, so are repeated interventions. These cells have been successfully used to generate osteogenic composite grafts with intrinsic vascularity in preclinical models.

For translation into clinical practice after a 20 patient external pilot a prospective randomized controlled trial with 270 patients is planned. For the trial lipoaspiration precedes open reduction and internal fixation in individuals over 60 years presenting with a proximal humeral fracture after low-energy trauma. Cells are isolated (Cellution®800/CRS) and wrapped around hydroxyapatite microgranules after embedding in a fibrin-gel for augmentation of the typical bone-void. Clinical/radiological follow-up is at 6 and 12 weeks for immediate complications and after 6, 9 and 12 months. Functional assessment is performed after 6 weeks, 6 and 12 months using the Quick-Dash- and Constant-Score.

The primary outcome is a reduction in secondary dislocation by 50% during the first postoperative year. Secondary dislocation is diagnosed on plain radiographs by an independent board certified radiologist specialised in musculoskeletal imaging if one or more of the following criteria are met:

* More than 20° varus collapse of the humeral head fragment in relation to the humeral shaft
* Screw penetration through the humeral head

ELIGIBILITY:
Inclusion Criteria:

Presentation with an isolated proximal humeral fracture after a low-energy trauma (e.g. falling from a standing position) and:

* indication for open reduction and internal fixation with a proximal humeral locking plate (PHILOS®, Synthes, Switzerland) after low energy trauma

  * displacement of more than 1 cm between fragments and/or
  * angulation of 45° or more between the fragments and/or
  * dislocation of the greater tuberosity of 5 mm or more and/or
  * patient specific factors like high functional demand etc
* age > 50 years
* postmenopausal status (i.e. 12 continuous month without menstruation)
* informed consent in surgery and study participation

Exclusion Criteria:

* Psychiatric disorder severely impairing co-operation (dementia mini mental Status (MMS) <24, schizophrenia, major depression)
* Pathological fractures caused by other conditions
* Fracture-related nerve injury
* Malignancies under current treatment (i.e. chemotherapy, radiotherapy etc.)
* BMI <20 kg/m2
* Known hypersensitivity to one of the graft components
* Participation in a clinical trial within 3 month before enrolment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Development of secondary dislocation within 12 months postoperative | 12 months postoperative
  Secondary dislocation within the first year postoperative on plain radiographs in ap. and Neer projections diagnosed by an independent radiologist specialized in musculoskeletal imaging in case of
  * more than 20° varus collapse of the humeral head fragment in relation to the humeral shaft
  * screw penetration through the humeral head

SECONDARY OUTCOMES:
Functional outcome 6 weeks, 6 and 12 months after fixation | 12 months postoperative
  Functional outcome 6 weeks, 6 and 12 months after fixation: the functional outcome will be recorded by the Quick Dash Score and the Constant at each follow up visit and compared between the two groups. Additionally, pain at either surgical site will be recorded via the visual analogue scale.
Safety | 12 months postoperative
  safety: all adverse reactions will be recorded and analysed to assess the safety of the approach in a typical patient population.
bone mineral density | 12 months postoperative
  bone mineral density: in case of implant removal (see below) a 100 mm3 bone biopsy will be taken from the grafted area and analysed with MicroCT (micro computed tomography) for bone mineral density.
Histology | 12 months postoperative
  histological assessment of qualitative and quantitative bone formation: bone biopsies will - after MicroCT assessment - be decalcified and histologically analysed using standard techniques and image quantification
Dose-response | 12 months postoperative
  establishment of a dose response relationship between number of implanted cells an bone quantity in microCT and histologically via image quantification: retrospectively the quantitative measures of bone formation will be correlated to the number of implanted cells and their clonogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Saxer, MD, Principal Investigator — University Hospital, Basel, Switzerland; Marcel Jakob, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196